CLINICAL TRIAL: NCT00298675
Title: A Phase 1/1b Dose Escalation Study Evaluating BSI-201 as a Single Agent and in Combination With Irinotecan in Subjects With Advanced Solid Tumors
Brief Title: Phase 1/1b Dose Escalation Study Evaluating BSI-201 as a Single Agent and in Combination With Irinotecan in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11483; 20060101 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — iniparib; Irinotecan

ARMS (2):
- Iniparib (Experimental)
  Interventions: Drug: BSI-201 (iniparib)
- Iniparib/irinotecan (Experimental)
  Interventions: Drug: BSI-201 (iniparib); Drug: irinotecan

INTERVENTIONS:
Drug: BSI-201 (iniparib) — BSI-201 administered intravenously (IV), 2x weekly
  Other Names: SAR240550
Drug: irinotecan — Irinotecan administered weekly, IV.
  Arms: Iniparib/irinotecan

SUMMARY:
The purpose of this study is to assess the safety, establish the maximum tolerated dose (MTD) and generate pharmacokinetic profiles of BSI-201 after IV administration in adult subjects with histologically documented advanced solid tumors that are refractory to standard therapy or for which no standard therapy is available. Additionally, the safety and tolerability and clinical response of BSI-201 + irinotecan will be investigated in patients with metastatic breast cancer in the phase 1b portion of the study.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, advanced solid tumor that is refractory to standard therapy or for which no standard therapy is available.
* ECOG performance status of 0, 1, or 2
* Adequate hematological status
* Any prior toxicity from prior chemotherapeutic treatment recovered to grade 1 or grade 0
* 18 years of age or older
* Competent to comprehend, sign, and date an Institutional Review Board (IRB) approved informed consent form
* For phase 1b portion only: metastatic breast cancer

Exclusion Criteria:

* Hematologic malignancies
* Symptomatic or untreated brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and corticosteroids
* Myocardial infarction within 6 months of study day 1, unstable angina, congestive heart failure with NYHA > class II, uncontrolled hypertension
* Known positive test for HIV or hepatitis C virus, or chronic active hepatitis
* Major surgery within 1 month of study day 1
* History of second neoplasm, except for curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix and other primary cancer with no known active disease present and no curative treatment administered for the last 3 years
* History of seizure disorder or currently on anti-seizure medication
* Systemic chemotherapy or radiation therapy within 28 days of study day 1
* Antibody therapy for treatment of underlying malignancy within 1 month of study day 1
* Evidence of liver disease shown by elevated enzymes
* Evidence of renal disease shown by serum creatinine > 1.5 x upper limit of normal
* Currently receiving platelet of GCF support for any medical condition
* Concurrent use of herbal medications taken with the intent to treat cancer
* Enrolled in or not yet completed at least 30 days since ending other investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | After one cycle

SECONDARY OUTCOMES:
Clinical Response | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Research Site, New Haven, Connecticut
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas